CLINICAL TRIAL: NCT02311179
Title: The Effect of Implant Coating With Hydroxyapatite Deposited Electrochemically (BoneMaster) on Migration and Clinical Outcome in Hip Arthroplasty With the Exceed Cup
Brief Title: The Effect of Implant Coating (BoneMaster) on Migration and Clinical Outcome in Hip Arthroplasty With the Exceed Cup
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Biomet Denmark Aps (Unknown); Project coordinator Orthopaedic Centre, Aarhus (Unknown); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20110224
Record Dates: First submitted 2012-11-06; First posted 2014-12-08 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis
Keywords: Prosthesis fixation; hip arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Prostheses and Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prosthesis, BoneMaster-Exceed cup (Active Comparator): Prosthesis, BoneMaster-Exceed cup: A hemispheric joint cup of the type Exceed cup (Biomet) characterized by a porous surface of titanium plasma spray. The surface is coated with hydroxyapatite deposited electrochemically (BoneMaster)
  Interventions: Device: Prosthesis, BoneMaster-Exceed cup (Biomet)
- Prosthesis Exceed cup without HA (Active Comparator): Prosthesis Exceed cup without HA: A hemispheric joint cup of the type Exceed cup (Biomet) characterized by a porous surface of titanium plasma spray
  Interventions: Device: Prosthesis Exceed cup without HA (Biomet)

INTERVENTIONS:
Device: Prosthesis, BoneMaster-Exceed cup (Biomet) — Patients will be randomized preoperatively to 1) Exceed cup coated with hydroxyapatite deposited electrochemically (BoneMaster) or 2) Exceed cup coated without hydroxyapatite coating.
  Arms: Prosthesis, BoneMaster-Exceed cup
Device: Prosthesis Exceed cup without HA (Biomet) — Patients will be randomized preoperatively to 1) Exceed cup coated with hydroxyapatite deposited electrochemically (BoneMaster) or 2) Exceed cup coated without hydroxyapatite coating.
  Arms: Prosthesis Exceed cup without HA

SUMMARY:
This study focuses on the effect of the hydroxyapatite coating with BoneMaster on the fixation of the hip prosthesis in primary hip alloplasty. A hemispheric joint cup of the type Exceed cup (Biomet) characterized by a porous surface of titanium plasma spray is used. The surface is coated with hydroxyapatite deposited electrochemically (BoneMaster) and will be compared with an identical cup without hydroxyapatite.

DETAILED DESCRIPTION:
This study focuses on the effect of the hydroxyapatite coating with BoneMaster on the fixation of the hip prosthesis in primary hip alloplasty. A hemispheric joint cup of the type Exceed cup (Biomet) characterized by a porous surface of titanium plasma spray is used. The surface is coated with hydroxyapatite deposited electrochemically (BoneMaster) and will be compared with an identical cup without hydroxyapatite. A 5-year radiologic analysis of migration will be carried out with the object of detecting prognostic evidence of prosthesis loosening. Migration is determined by Roentgen Stereo-photogrammetric Analysis (RSA) on stereoroentgenography. Simultaneously, the patients will be monitored by using the clinical outcome measure HOOS (Hip disability and osteoarthritis outcome score), OHS (Oxford Hip Score), EQ-5D (EuroQol), HHS (Harris Hip Score) on range of motion, VAS (Visual Analog Scale), postoperative complications and reoperation.

Hypothesis: We expect that the Exceed cup with hydroxyapatite deposited electrochemically (BoneMaster) is superior or equal compared to a similar cup without hydroxyapatite regarding

* mechanical stability (RSA)
* (clinical outcome)

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic radiographic osteoarthritis
2. Radiographically and clinically adequate bone quality with regard to a total hip prosthesis, including osteoporosis-Dexa-Scanning verification.
3. Age 55 to 75 years
4. Informed written consent

Exclusion Criteria:

Orthopaedic

1. Other disease of affected hip than primary coxarthrosis at time of inclusion 1.1. Secondary osteoarthritis 1.1.1. sequelae after acetabular fracture 1.1.2. hip-near femoral fracture 1.1.3. calve perthe 1.1.4. dysplasia (severe) 1.1.5. other 1.2 Atraumatic caput necrosis
2. Neuromuscular or vascular condition in one or the other lower extremity
3. Immobilization postoperative for long periods, for instance because of other serious diseases, alloplasties of the other lower-extremity joint, etc (decided by investigator)
4. Reoperation of affected hip because of 4.1 luxation (with closed or open reduction) 4.2 deep infection 4.3 fracture 4.4 aseptic loosening 4.5 other
5. Body Mass Index (BMI) at time of inclusion 81-84 5.1 ≥ 35 kg/m2 (grade 2+3 85, Obese Class I 81) 5.2 < 18,5 kg/m2 81-84
6. Insufficient RSA marker spread or rigidity Operative
7. Use of component other than Bimetric femoral stem (HA porous-coated without collar)
8. Unsuitable bone quality for uncemented hip alloplasty, evaluated preoperatively
9. Complications peroperatively on insertion of hip alloplasty that necessitate deviation for the described operative procedure (see section: "Operative procedure"), among others 9.1 per- and postoperative fracture 9.2 bone graft used peroperatively (treatment of bone defects, cysts, etc.) 9.3 screw fixation of the acetabulum 9.4 gluteal detachment or extensive femoral exposure 9.5 trochanter osteotomy 9.6 Under-reaming 1-2 mm (cup size is one mm larger than the reamer, i.e. reaming 51 mm, cup 52 mm) 9.7 Other Radiographic
10. Cup placement 10.1 Cup inclination in AP (anteroposterior) plan >56 degrees and <35 degrees as evaluated on roentgenogram Medical
11. Osteoporosis 11.1. previously diagnosed 11.2. project-related preoperative DEXA (dual energy x-ray absorptiometry ) scan Patients with osteoporosis on the scan (T-score < -2.5) are excluded from the study with referral to medical osteoporosis treatment. Patients with osteopenia (T-score < -1) are included in the project with referral to osteoporosis prophylactic treatment. Patients with osteopenia at project inclusion are DEXA re-scanned at the 2 year follow up.
12. Arthritis 12.1. rheumatoid arthritis 12.2. psoriasis arthritis 12.3. other arthritides
13. Metabolic bone disease 13.1. hyperparathyroidism 13.2. Paget bone disease 13.3. renal osteodystrophy 13.4. other
14. Reduced kidney function thereby influencing bone metabolism
15. Previous treatment of skeleton with radiation therapy
16. Cancer Pharmaceuticals
17. Pharmaceuticals that effect calcium-phosphorus metabolism and bone density 87-98, either through intermittent administration or as a constant dose 17.1. glucocorticoids (systemic) beyond short-term treatment (<5 days) 17.2. immunosuppression/modulation (cyclosporine, methotrexate, etc.) Compliance related
18. Absent patient compliance with treatment and follow-up investigations
19. Abuse that the investigator feels would weaken compliance 19.1. alcohol abuse 19.2. medication abuse
20. Psychological instability (including patient in treatment lithium/antidepressants/neuroleptics/ antipsychotic drugs) which the investigator feels would weaken compliance

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Radiographic: Migration of the acetabular component (mm, degree) with Model-Based RSA (m-RSA) | End of study (up to 5 years)

SECONDARY OUTCOMES:
Reoperation of affected hips | End of study (up to 5 years)
Postoperative complications (up to 5 years) | End of study
HOOS (Hip disability and osteoarthritis outcome score) | End of study (up to 5 years)
OHS (Oxford Hip Score) | End of study (up to 5 years)
HHS (Harris Hip Score) on Range Of Motion (ROM) | End of study (up to 5 years)
VAS (Visual Analog Scale) at rest and load | End of study (up to 5 years)
EQ-5D (EuroQol) | End of study (up to 5 years)
Radiologic osteolysis | End of study (up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, Prof, dr med, Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Jorgensen PB, Krag-Nielsen N, Lindgren L, Morup RMS, Kaptein B, Stilling M. Radiostereometric analysis: comparison of radiation dose and precision in digital and computed radiography. Arch Orthop Trauma Surg. 2023 Sep;143(9):5919-5926. doi: 10.1007/s00402-022-04674-0. Epub 2022 Nov 23. PMID 36422666